CLINICAL TRIAL: NCT03415711
Title: A Double-blind, Randomized, Placebo-controlled, Single-center, Dose-finding, Pilot Study Evaluating the Efficacy of VSL#3® in the Maintenance of Clinical and Endoscopic Remission of Mild-to-moderate UC
Brief Title: PRObiotic VSL#3® for Maintenance of Clinical and Endoscopic REMission in Ulcerative Colitis
Acronym: PROREM UC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: VSL Pharmaceuticals (Industry)
Collaborators: Actial Farmaceutica S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDIVSL01
Record Dates: First submitted 2018-01-05; First posted 2018-01-30 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mesalamine plus high-probiotic preparation VSL#3® (Experimental): Mesalamine 2.4 g/day in once daily administration plus VSL#3® 450 billion sachets, two sachets per day (900 billion of bacteria per day) for 12 months.
  Interventions: Dietary Supplement: VSL#3®; Drug: Mesalamine
- Mesalamine plus low-probiotic preparation VSL#3® (Experimental): Mesalamine 2.4 g/day in once daily administration plus VSL#3® 450 billion sachets, two sachets twice a day (1800 billion of bacteria per day) for 12 months.
  Interventions: Dietary Supplement: VSL#3®; Drug: Mesalamine
- Mesalamine plus Placebo (Active Comparator): Mesalamine 2.4 g/day in once daily administration plus placebo for 12 months.
  Interventions: Drug: Mesalamine; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3® — VSL#3® 450 billion sachets
  Arms: Mesalamine plus high-probiotic preparation VSL#3®; Mesalamine plus low-probiotic preparation VSL#3®
Drug: Mesalamine — Mesalamine 2.4 g/day in once daily administration.
Drug: Placebo — sachets with maltose, cornstarch and dioxide
  Other Names: Placebo (for VSL#3®)
  Arms: Mesalamine plus Placebo

SUMMARY:
Ulcerative colitis (UC) is an inflammatory bowel disease (IBD) characterized by chronic inflammation limited to colonic mucosa. Its pathogenesis is not still clear, even if a multifactorial aetiology has been advocated. The aim of this study is to evaluate the long-term efficacy of two different doses of VSL#3® added on standard therapy (5-ASA) in maintaining remission in an adult population of patients with UC, compared with the standard therapy (5-ASA) plus placebo. The investigators hypothesized that adding VSL#3® to mesalamine would lead to higher remission rate at long-term evaluation.

DETAILED DESCRIPTION:
This is a Phase II a, parallel-groups, randomized, double-blind, placebo-controlled, single-center, dose finding study in subjects with UC in remission. Two different oral doses of VSL#3® added to standard therapy (5-ASA) will be investigated compared to standard therapy (5-ASA) plus placebo (in a 1:1:1 ratio).

All patients will receive standard therapy for maintaining remission. 39 subjects will be randomly assigned to 1 of the 3 treatment arms for the 12-month treatment period as following:

* group A: 13 patients will receive mesalamine 2.4 g/day in once daily administration plus VSL#3® 450 billion sachet, two sachets per day for 12 months (900 billion of bacteria per day)
* group B: 13 patients will receive mesalamine 2.4 g/day in once daily administration plus VSL#3® 450 billion sachet, two sachets twice a day (1800 billion of bacteria per day) for 12 months
* group C: 13 patients will receive mesalamine 2.4 g/day in once daily administration plus placebo for 12 months.

Subject participation in this study will be approximately 20 months which includes up to a 8-week screening period, a 12-month treatment period, and a 6-month follow-up period. At the conclusion of the 12-month treatment period, subjects will continue in the 6-month follow-up period (telephone contact conducted after 6 months).

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
2. Subjects are willing and able to participate in the study, complete subject assessments, attend scheduled clinic visits, and comply with all protocol requirements as evidenced by written informed consent.
3. Male and/or female subjects aged ≥18 years at the time of informed consent.
4. A diagnosis of UC for ≥3 months. A biopsy report must be available to confirm the histological diagnosis in the subject's source documentation. In addition, a report documenting disease duration and extent of disease (e.g., proctosigmoiditis, left-sided colitis and pancolitis) based upon prior colonoscopy must also be available in source documentation.
5. Must have a flexible sigmoidoscopy indicative of UC in remission (Mayo endoscopic subscore ≤1) during screening period, to be performed after all other inclusion criteria have been met.
6. Must have history of previous mild-to-moderate active disease beyond the rectum (>15 cm from the anal verge).
7. Must have UC in remission with a Total Mayo Score ≤2 with no individual subscore>1 and rectal bleed subscore of 0.
8. Must be on maintenance treatment with oral mesalamine (<2.5 g/day), sulfasalazine (<3.0 g/day) or olsalazine (<1.5 g/day) on a stable dose for at least 2 weeks before randomization.
9. Male and female subjects of childbearing potential must agree to avoid pregnancy throughout the duration of the study (defined as the time of the signing of the informed consent through the conclusion of subject participation). A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.

   * Women of childbearing potential (WOCBP) must have a negative urine pregnancy test result at screening. WOCBP are defined as women who are biologically capable of becoming pregnant, including women who are using contraceptives or whose sexual partners are either sterile or using contraceptives.
   * Women of non-childbearing potential (WONCBP) do not require a urine pregnancy test and must meet at least one of the following criteria:

     * Have undergone hysterectomy or bilateral oophorectomy;
     * Have medically confirmed ovarian failure or are medically confirmed to be post-menopausal (cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; laboratory confirmation of Follicle-stimulating hormone (FSH) level may be indicated if subject has history of amenorrhea for ≥ 52 weeks).
     * Are medically confirmed to be post-menopausal (cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; laboratory confirmation of FSH level may be indicated if subject has history of amenorrhea for ≥ 52 weeks).

Exclusion Criteria:

1. Subjects with a diagnosis of indeterminate colitis or Crohn's disease. Subjects with clinical findings suggestive of Crohn's disease, e.g., fistulae or granulomas on biopsy are also excluded.
2. Subjects with colonic dysplasia or neoplasia.
3. Subjects with a history of colonic or small bowel obstruction or resection, except for appendectomy.
4. Use of rectal 5-aminosalicylic acid or systemic or rectal corticosteroids within 30 days before baseline, use of immunosuppressive agents within 12 weeks before baseline.
5. Use of antitumor necrosis factor (anti-TNFα) or anti-integrin therapy for UC at any moment of previous patient history 6. Repeated use of non-steroidal anti-inflammatory drugs (NSAIDs), including the non-steroidal anti-inflammatory drugs such as aspirin or ibuprofen (except for prophylactic use of a stable dose of aspirin up to 325 mg / day for cardiac disease). Occasional use of NSAIDs is permitted.

8. Subjects who had received another investigational agent within 30 days before baseline.

9. Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, immunologic, or local active infection/infectious illness) that, in the investigator's judgement will substantially increase the risk to the subject if he or she participates in the study.

10. Women during pregnancy or lactation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
To characterize the efficacy of VSL#3® plus standard therapy (5-ASA) in maintaining clinical and endoscopic remission in patients with UC in remission. | 12 months
  Proportion of subjects in clinical and endoscopic remission at month 12 as defined by Total Mayo Score ≤2 with no individual subscore>1 and rectal bleed subscore of 0.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Armuzzi, Principal Investigator — Policlinico Universitario Agostino Gemelli Università Cattolica del Sacro Cuore
Locations (1):
- Istituto di Medicina Interna CIC Columbus Policlinico Universitario Agostino Gemelli Università Cattolica del Sacro Cuore, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided